CLINICAL TRIAL: NCT04278482
Title: "Diseño y Validación en Humanos de un Nuevo Complemento Alimenticio Rico en Ácido Docosahexaenoico (DHA) Procedente de Algas"
Brief Title: Effects of the Consumption of a Supplement Rich in Docosahexaenoic Acid (DHA) From Algae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Comunidad de Madrid (Other)
Responsible Party: Principal Investigator, M Pilar Vaquero, Dr, National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: IND2018/BIO-9554
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Vegetarian Diet
Keywords: Vegetarian diets; Plant-based diets; Vegetarians; Vegans; docosahexaenoic acid; DHA; omega-3 fatty acids; algae; supplementation
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DHA supplement (Active Comparator): Supplement rich in DHA form algae source
  Interventions: Dietary Supplement: Dietary supplement, DHA or Placebo
- Placebo (Placebo Comparator): Placebo supplement
  Interventions: Dietary Supplement: Dietary supplement, DHA or Placebo

INTERVENTIONS:
Dietary Supplement: Dietary supplement, DHA or Placebo — Consumption of 2 capsules per day of the dietary supplement, DHA or Placebo

SUMMARY:
Vegetarian diets are increasing worldwide. To prevent nutritional deficiencies, supplementation with nutrients that are only present in animal food can be needed. In relation to fatty acids, vegetarian diets involve low intake of omega-3 polyunsaturated fatty acids (n-3 PUFA) and low blood levels of the long-chain n-3 derivatives, whose main dietary sources are fish and shellfish, particularly the levels of docosahexaenoic acid (DHA), which has important health benefits, are low.

In this regard, validation of supplements rich in the n-3 fatty acid DHA that are not obtained from fish is needed, thus the study will test the bioavailability and metabolic effects of a DHA supplement form algae.

The study will be conducted on the effects of the DHA supplement versus placebo in vegetarian and non-vegetarian healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥18 and ≤45 years).
* Healthy.
* Women.
* Men.
* Participant following either a vegetarian diet during at least 6 months or following a omnivorous diet but consuming fish 2 times per week or less.

Exclusion Criteria:

* Age <18 and >45 years old.
* Pregnancy.
* Diseases: liver diseases, gastric diseases, irritable bowel, hypercholesterolemia, hypertension, diabetes, biliary colic.
* Having participated in a clinical study in the last 3 months.
* Eating disorders.
* Consumption of foods fortified with omega-3 fatty acids in the last 3 months.
* Consumption of supplements of omega-3 fatty acids in the last 3 months.
* Participant who have followed either a vegetarian diet for less than six months or an omnivorous diet including fish more than 2 times per week.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Serum DHA | Baseline
  Docosahexanoic acid concentration in serum
Serum DHA | week 6
  Docosahexanoic acid concentration in serum
Serum DHA | week 12
  Docosahexanoic acid concentration in serum
Serum DHA | week 18
  Docosahexanoic acid concentration in serum

CONTACTS AND LOCATIONS:
Overall Officials: M.Pilar Vaquero, Dr, Principal Investigator — CSIC
Locations (1):
- M.Pilar Vaquero, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garcia-Maldonado E, Alcorta A, Zapatera B, Vaquero MP. Changes in fatty acid levels after consumption of a novel docosahexaenoic supplement from algae: a crossover randomized controlled trial in omnivorous, lacto-ovo vegetarians and vegans. Eur J Nutr. 2023 Jun;62(4):1691-1705. doi: 10.1007/s00394-022-03050-3. Epub 2022 Nov 23. PMID 36418565